CLINICAL TRIAL: NCT00125892
Title: A 1-Year Safety Study of Duloxetine in Patients With Fibromyalgia Syndrome
Brief Title: A Study of Duloxetine in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9075; F1J-MC-HMEH
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine

SUMMARY:
This study is designed to evaluate duloxetine for the treatment of fibromyalgia syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for primary fibromyalgia syndrome as defined by the American College of Rheumatologists

Exclusion Criteria:

* Treatment with a monoamine oxidase inhibitor within 14 days prior to Visit 2 or the potential need to take within 5 days after discontinuation from the study.
* Any patients judged by their physicians to be at serious suicidal risk.
* Have uncontrolled narrow-angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2005-07; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and efficacy of duloxetine in patients diagnosed with fibromyalgia syndrome

SECONDARY OUTCOMES:
Evaluate persistence of efficacy
Evaluate long-term differences in efficacy in different doses
Evaluate gains in efficacy in non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Capital Federal
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Cotton Tree, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Malvern, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Hobart
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Melbourne
- Brazil (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Recife
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, São Paulo
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, St. John's, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Saskatoon, Saskatchewan
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Morelia, Michoacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Mérida, Yucatán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday -Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday -Friday from 9:00AM to 5:00PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Mexico City
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Lublin
  - For additional information regarding investigative sites for this trial. contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Wroclaw
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00PM Eastern Time (UTC/GMT - 5 hours , EST) or speak with your personal physician, Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your person physician, Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours , EST ) or speak with your personal physician, Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Taoyuan District

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com